CLINICAL TRIAL: NCT03955406
Title: Comparison of Low Flow Anesthesia With and Without Initial High Flow Phase
Brief Title: Low Flow Anesthesia Without Initial High Flow Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, MAHMUT ARSLAN, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KSU 2017-15
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Low Flow Anesthesia; Volatile Anesthetic Consumption

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): After standart intravenous anesthesia induction end endotracheal intubation desflurane vaporizer will be set at 6% with fresh gas flow rate 4 L/min (50% O2, 50% air) until the EtAA concentration reaches 0.7 MAC (minimum alveolar concentration) Then, the desflurane vaporizer will be at a 1% higher value than the EtAA concentration required to achieve 0.7 MAC. And after 10 minutes fresh gas flow rate will be reduced to 1L/min.
  Interventions: Procedure: Conventional Low flow Anesthesia
- Fixed Fresh Gas Flow Rate group (Active Comparator): After standart intravenous anesthesia induction end endotracheal intubation desflurane vaporizer will be set at 18% with fresh gas flow rate 1 L/min (50% O2, 50% air) until the EtAA concentration reaches 0.7 MAC (minimum alveolar concentration) Then, the desflurane vaporizer will be at a 2% higher value than the EtAA concentration required to achieve 0.7 MAC.
  Interventions: Procedure: Low Flow Anesthesia with fixed fresh gas flow rate

INTERVENTIONS:
Procedure: Conventional Low flow Anesthesia — During the initial wash-in period 4 L/min Fresh gas flow will be used.
  Arms: Conventional group
Procedure: Low Flow Anesthesia with fixed fresh gas flow rate — Fresh gas flow rate will be 1 L/min throughout the procedure.
  Arms: Fixed Fresh Gas Flow Rate group

SUMMARY:
The aim of the study is to compare the effectiveness of conventional low flow anesthesia (LFA) with initial high fresh gas flow ( 4L/min) for 10 minutes and LFA with fixed fresh gas flow rate (1L/min).

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* scheduled for surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* hemodynamic instability
* emergency cases
* expected anesthesia duration < 60 min
* patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
The time required to reach 0.7 MAC | perioperative
number of adjustments made to the vaporizer settings | perioperative
  MAC will be held between 0.6-0.8 with adjustments at the vaporizer

SECONDARY OUTCOMES:
anesthetic agent consumption | perioperative
  desfluane consumption at the first hour and at the end of the surgery wil be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://link.springer.com/article/10.1007%2Fs10877-018-0135-2